CLINICAL TRIAL: NCT01495377
Title: Does Opioid Induced Swallowing Difficulty Lead to Elevated Risk for Pulmonary Aspiration?
Brief Title: Opioid Induced Swallowing Difficulties and Risk for Pulmonary Aspiration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Johanna Savilampi, principal investigator, Region Örebro County
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JS003
Record Dates: First submitted 2011-12-09; First posted 2011-12-20 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Opioid Induced Swallowing Disorders
Keywords: swallowing difficulties; remifentanil; pulmonary aspiration; scintigraphy
MeSH Terms: conditions — Deglutition Disorders | interventions — Remifentanil; Sodium Chloride; Technetium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Remifentanil (Active Comparator)
  Interventions: Drug: Remifentanil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Technetium (Experimental)
  Interventions: Drug: Technetium
- Dynamometer (Experimental)
  Interventions: Device: Dynamometer (Jamar)

INTERVENTIONS:
Drug: Remifentanil — Powder for injection/ infusion fluid solution, 1 mg Infusion TCI 3 ng/ml 60 min ( 0,15 ug/kg/min)
  Other Names: Ultiva; ATC-code: N01AH06
  Arms: Remifentanil
Drug: Placebo — Infusion fluid, solution 9 mg/ml ( hydrogenic solution )
  Other Names: Saline; ACT-code: B05XA03
  Arms: Placebo
Drug: Technetium — 37-40 MBq( effective dose 0,7 mSv) 99Tc albumin colloid in a volume of 6 ml, infusion velocity 0,1 ml/min via a transnasal catheter
  Other Names: Nanocol; ACT-code: V09DB01
  Arms: Technetium
Device: Dynamometer (Jamar) — portable hydraulic hand dynamometer to assess grip strength.
  Other Names: Jamar dynamometer
  Arms: Dynamometer

SUMMARY:
The purpose of this study is to determine weather remifentanil induced swallowing difficulties increase risk for pulmonary aspiration.

DETAILED DESCRIPTION:
Remifentanil and other opioids are widely used as anesthetic sedation during minor surgical procedures and as pain relief in icu-patients when the patient is spontaneously breathing and the airway is not secured by endotracheal intubation. In these circumstances inability to clear the pharynx by swallowing may increase risk for aspiration.In a previous study ( not yet published) we showed that remifentanil induce subjective swallowing difficulties in healthy volunteers and the aim of this study is to determine weather remifentanil infusion in healthy non-intubated volunteers increase risk for pulmonary aspiration. To assess this question we are going to study 14 volunteers who are randomised to receive remifentanil infusion with target concentration 3 ng/ml during 60 minutes at one occasion and an equal amount of saline at the other. Radioactive Technetium colloid solution is parallelly infused through a pliable catheter transnasally. After remifentanil infusion is stopped the transnasal catheter is removed and the volunteer is asked to swallow water to clear the remaining radioactivity from upper gastrointestinal tract. Thereafter lung scanning with a gamma camera is performed. Through which mechanism remifentanil cause swallowing difficulties is not known.To determine weather remifentanil induce general muscle weakness in volunteers measurements of grip strength using Jamar dynamometer are performed before, during and 15 minutes after remifentanil infusion.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 year old healthy volunteers from both sexes.
* Have signed and dated Informed Consent.
* Willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

* Pharyngoesophageal dysfunction
* Anamnesis of pharyngoesophageal dysfunction
* Known history of cardiac, pulmonary or neurological disease
* Ongoing medication
* Allergies to or history of reaction to naloxone, remifentanil, fentanyl analogues or other ingredients
* History of reaction to products containing human albumine
* Pregnancy or breast feeding
* BMI > 30
* Previous participation in a medical clinical trial where opioid has been used or have during last 30 days participated in any other medicinal clinical trial or in a trial where follow-up in not completed

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Radioactivity evident in lungs imaged using a gamma camera | one study occasion takes two hours and a gamma camera scan is taken in the end of the occasion

SECONDARY OUTCOMES:
Grip strength measured with Jamar dynamometer | volunteers are studied during two hours during which grip strength is measured three times
  Jamar dynamometer is positioned in the dominant hand att maximal grip strength contraction is taken three times, the mean value is used for the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: magnus wattwil, MD, PhD, Study Chair — University Hospital in Örebro
Locations (2):
- Sweden (2):
  - University Hospital in Örebro, Örebro
  - Örebro University Hospital, Örebro